CLINICAL TRIAL: NCT00732680
Title: Prospective Case Series Evaluating Short and Long Term Benefits of the Use of Botox in the Treatment of Empty Nose Syndrome
Brief Title: Benefits of the Use of Botox in the Treatment of Empty Nose Syndrome Syndrome
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lead investigator moved to a new medical center; study was stopped when he left.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-005015
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Empty Nose Syndrome; Atrophic Rhinitis
Keywords: Empty nose syndrome; Over resection of turbinate; Atrophic rhinitis
MeSH Terms: conditions — Rhinitis, Atrophic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botulinum Toxin Type A (Experimental): Treatment will be in the form of 10 Units of Botulinum Toxin Type A injected into the dilator nasalis muscle on each side of the nose.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 10 Units of Botulinum Toxin Type A injected into the dilator nasalis muscle on each side of the nose.
  Other Names: Botox

SUMMARY:
Empty Nose Syndrome patients suffer from disabling physical symptoms and considerable distress. To date there is no definitive cure for these symptoms. Established treatment modalities include saline irrigation, surgical implantation of materials or simply use of cotton wads/ silicon cones to simulate the resistive action to airflow of the resected turbinates.

This study will research the effectiveness of a new treatment modality in the treatment of Empty Nose Syndrome. This novel treatment method involves the use of botulinum toxin type A (Botox).

DETAILED DESCRIPTION:
Background:

Empty Nose Syndrome (ENS) is the term used to describe the condition resulting from over resection of nasal turbinate. Symptoms include depression, dysosmia, bleeding, discharge, crusting, dryness, dysosmia, and pain.

Treatment modalities include adjunctive comfort measures (primarily irrigation), mechanical measures (Silicon cones, cotton wads) and surgical treatment (alloderm implants, plastipore cartilage grafts etc.) We will investigate a new method of treatment for ENS. This will involve injection of botulinum toxin type A into the dilator nasalis muscle thus collapsing the internal nasal valve to provide added resistance to air flow.

Objective:

To evaluate effectiveness of botulinum toxin type A in improving overall quality of life in ENS patients.

Methods:

ENS patients in this study will receive botulinum toxin type A along with adjunctive treatment which will include several measures. First of all, patients will be given a nasal rinse bottle and will be instructed to irrigate their noses twice a day as follows:

* Irrigate the nose 250cc (about 125cc each side) to clear the mucus.
* Stop and gently clear the nose.
* Irrigate the nose 250cc (about 125cc each side) once again.
* Sit quietly for 10 minutes. No blowing.
* Do not blow the nose for 2 hours.

Patients will be asked to use sesame oil once a day to prevent drying of the nasal mucosa with further administration as needed. In addition they will advised to make certain lifestyle modifications that will include sleeping with a cool mist humidifier, drinking plenty of fluids and engaging in regular physical activity.

Before and after treatment data will be obtained in the form of a breathing test and patient questionnaires that will measure changes in physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 18-65 years of age presenting with a known diagnosis of ENS who has no known allergies to Botox.

Exclusion Criteria:

* Patients younger than 18 years or older than 65 years of age.
* Patients with neuromuscular disorders or neuropathic diseases.
* Patients with infection and or swelling at the site where Botox is to be injected.
* Patients with known hypersensitivity to any ingredient in the drug formulation (botulinum toxin, human albumin)
* Patients who are or plan to become pregnant within the time period in which the study will be conducted.
* Patients who are nursing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oren Friedman, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Online listing of the study with study details and contact information. — http://www.clinicaltrials.gov
- See also: FDA website. Great website for information on Botox. — http://www.fda.gov/
- See also: online blog of people with empty nose syndrome. — http://www.emptynosesyndrome.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botulinum Toxin Type A
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Score of Sino Nasal Outcome Test 22 (SNOT 22)
Description: The SNOT 22 is a validated measure of health related quality of life in sinonasal disease. It is a 22 item questionnaire with each item assigned a score ranging from 0-5. The total score may range from 0-110 and lower scores represent better health related quality of life.
Time Frame: 2 weeks after intervention, 2 months
Population: No study data was collected in the study. The Lead investigator moved to a new medical center; the study was stopped when he left.
Arm/Group | Botulinum Toxin Type A
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin Type A
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

LIMITATIONS AND CAVEATS:
No study data was collected in the study. The Lead investigator moved to a new medical center; the study was stopped when he left.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No